CLINICAL TRIAL: NCT04329663
Title: Effectiveness of the Indonesian Computer-based Game Prototype Towards ADHD Clinical Symptoms and Executive Function: A Functional Magnetic Resonance Imaging-blood-oxygen-level-dependent Pilot Study
Brief Title: Effectiveness of the Indonesian Computer-based Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tjhin Wiguna (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other); Fakultas Kedokteran Universitas Indonesia (Other); Binus University International (Unknown)
Responsible Party: Sponsor-Investigator, Tjhin Wiguna, Prof. Dr. dr., Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Indonesian computer-based game
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: ADHD; Executive Function
Keywords: Indonesia, computer-based game; executive function; ADHD; BRIEF; CATPRS; Primary school children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The inclusion criteria was child with ADHD age 5 to 12 years old that never taken medication prior to the study and willing to undergo training with computer based game which developed from phase one of the study for about 20 sessions with approximately 30 minutes per each session for 4 weeks consecutively. The training was conducted at school where the sample attended school so it would not disturb the learning and teaching process at school. The training would be guided and supervised directly by the researcher team.
  The diagnosis of ADHD was conducted by trained child and adolescent psychiatrist guided by Mini-Kids which was structured interview guide built based on ICD-X. Children which included on the study were child with ADHD without any other mental disorder comorbidity and does not has chronic physical illness during the interview with the parents. Child which does not complete 90% of the numbers of the training that planned will not included in data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- training group (Experimental): Ten children with ADHD who got the 20 sessions training of the Indonesian computer-based game prototype. They we were assessed by CATPRS, BRIEF and fMRI BOLD
  Interventions: Device: Indonesian computer-based game prototype

INTERVENTIONS:
Device: Indonesian computer-based game prototype — In order to improve the ADHD clinical symptoms and executive function of the player, this game should has challenge similar to memory game which is the player was given object to be memorized and then match the object in accordance to the task given inside the game. With some difficulty leves, this game was tried to trigger players in terms of accuracy and quickness in completing the mission.

SUMMARY:
The aim of this study was to develop an Indonesian computer-based game prototype that targets the clinical symptoms of ADHD as well as executive function and to investigate effectiveness through fMRI BOLD examination. This was a mix-method study design; the first step was an exploratory qualitative study using focused group discussion. The second step was 'the one group pre- and post-test design study' without any control. Ten primary school children who were drug-naïve and had a diagnosis of ADHD with no other mental or physical disorders participated in the study. Clinical improvement was measured by the CATPRS, BRIEF, and fMRI BOLD examination that focused on DLPFC-Hippocampus functional connectivity before and after 20 sessions of the Indonesian computer-based game prototype training. Data were analyzed using the paired t test and Pearson's correlation in SPSS for Mac version 21, and fMRI BOLD functional analysis was performed using SPM software version 12 and CONN Toolbox version 17. The hypothesis was: the Indonesian computer-based game prototype had an effect towards ADHD clinical symptoms and executive function that correlated with DLPFC-Hippocampus functional connectivity.

DETAILED DESCRIPTION:
This study had two phases and was designed as a mix-method study. The first step was an exploratory qualitative study, and the second was a quasi-experimental study without any control.

1. First Phase On the first phase, study conducted by using qualitative explorative design to develop and create computer-based game with Indonesian content in order to increase working memory capacity. This phase was done by focus group discussion (FGD) approach which involve participation from Indonesian Game Laboratorium from Faculty of Computer Science of Binus University International; and child and adolescent psychiatrist from Department of Psychiatry dr Cipto Mangunkusumo General Hospital - Faculty of Medicine Universitas Indonesia, Jakarta. .
2. Second Phase:

On the second phase of the study, it used ' the one group pre- and post-test' without control design which aims to prove that the predeveloped game has impact to executive function of the child and impact to DLPFC region of the brain. The inclusion criteria was child with ADHD age 5 to 12 years old that never taken medication prior to the study and willing to undergo training with computer based game which developed from phase one of the study for about 20 sessions with approximately 30 minutes per each session for 4 weeks consecutively. The training was conducted at school where the sample attended school so it would not disturb the learning and teaching process at school. The training would be guided and supervised directly by the researcher team.

The diagnosis of ADHD was conducted by trained child and adolescent psychiatrist guided by Mini-Kids which was structured interview guide built based on ICD-X. Children which included on the study were child with ADHD without any other mental disorder comorbidity and does not has chronic physical illness during the interview with the parents. Child which does not complete 90% of the numbers of the training that planned will not included in data analysis. Number of study's subject which needed on this research was obtained by using sample size table formula for clinical studies', with α = 0,05, β=0,2, 2-sided and consider that Δ (effect size) = 1 resulting that 10 subjects were needed. This formula was used because to date, similar study has not found or conducted ( training with game and imaging with fMRI BOLD)

Operational definition which used in this study are:

1. ADHD (Attetion Deficit Hyperactivity Disorder) defines as neurodevelopmental disorder which marked by hyperactivity, impulsive behaviour and difficulty in concentrate which happens more often and severe compares to peer group from same age group. This disorder causes impairment and distress to the child and his/her family. Diagnosis of ADHD and exclusion of other mental disorder was conducted by trained child and adolescent psychiatrist which established by structured interview using MINI kids.
2. Working memory deficit defines as deficit in ability to store and manipulate information for a short period of time and to be able to look upon, memorize, and take action on an information simultaneously. Clinical measuring of working memory deficit is done by BRIEF questionnaire which have been validated into Indonesion language 2011.
3. Imaging with fMRI was conducted by special stimuli to stimulate child's executive function with go and no-go modification which were images that had to be memorized in accordance to specific order and truth of the image. fMRI was conducted at Radiology Unit, Abdi Waluyo Hospital, using MRI scanner from GE Health care, 3 Tesla, 8-channel-coil. Sequence which used was Echo Plannar Imaging (EPI), with some modification; TR 3 seconds, TE 30, bandwidth 250kHZ, FOV 240 x 240, slice thickness 3 mm, space 1 mm, matrix 84 x 84 (frequency x phase), NEX 1, total slices 36, time 312 seconds. The measuring would be changes in activity by imaging result of fMRI BOLD (blod Oxygen-Level Dependent Contrast), which the level will increase on the more active brain part and decrease on the less active brain part.

Data Analysis Qualitative data was analysed by qualitative approach and described in a form of text. Data analysis for quantitative study was conducted by 't' test analytic for variable dependent by SPSS version 21 for Mac.

Data from MRI result would undergo pre-processing process which are realignment, writing and smoothing with FHWM 8 mm, then processed with Statistical Parametric Mapping (SPM) software version 12 and CONN Toolbox version 17. Analysis method which conducted was ROI-to ROI method wth the chosen ROI for this studty were lef and right Dorsolateral Prefrontal Cortex and Hippocampus fucntional connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Children with ADHD diagnosis
* Aged 6 to 12 years who were drug-naïve prior to the study, does not have any other mental or physical chronic illnesses, and willing to undergo the Indonesian computer-based game prototype training for 20 sessions with approximately 30 minutes per session over 4 weeks consecutively

Exclusion Criteria:

* N/A

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
ADHD clinical symtpoms-parent rating | 5 - 10 minutes
  Connors' Abbreviated Parent Teacher Rating Scale. The total lower score lower score is 0 and the higher total score is 30
ADHD clinical symtpoms-teacher rating. The total lower score lower score is 0 and the higher total score is 30 | 5 - 10 minutes
  Connors' Abbreviated Parent Teacher Rating Scale
executive function | 15 - 20 minutes
  Behavior Rating Inventory of Executive Function (BRIEF). The raw data is transformed into the Tscore. The anaylsis using the Tscore
DLPFC-Hippocampus functional connectivity | 20 - 30 minutes
  functional Magnetic Resonance Imaging Brain Oxygen Dependent Level. The functional connectivity is generated from the Conn toolsbox ans SPM 12.

CONTACTS AND LOCATIONS:
Overall Officials: Tjhin Wiguna, PhD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital; Tjhin Wiguna, PhD, Principal Investigator — Fakultas Kedokteran Univeristas Indonesia
Locations (1):
- dr. Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Study protocol